CLINICAL TRIAL: NCT01251029
Title: Ability of N-acetylcysteine to Prevent Deterioration in Renal Functioning in CKD Patients Undergoing Major Surgery Under General Anesthesia
Brief Title: Effect of N-acetylcysteine on Renal Functioning of Chronic Kidney Diseases(CKD) Patients After General Anesthesia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Dr. Bahar Murat, MD, Anesthesiology Department, Assaf Harofeh Medical Center
Other Study IDs: 197/10
Record Dates: First submitted 2010-11-25; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Kidney Diseases; General Anesthesia
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Acetylcysteine

ARMS (1):
- sugar pil and saline (Experimental)
  Interventions: Drug: N-acetylcysteine; Drug: Siran (N-acetylcysteine)

INTERVENTIONS:
Drug: N-acetylcysteine — 1200 mg orally; 600mg i.v.
Drug: Siran (N-acetylcysteine)

SUMMARY:
Acute kidney injury (AKI) is one of the most serious and frequent complication of general anesthesia. Patients suffer from chronic kidney diseases (CKD) predispose to develop AKI. CKD patients often need some surgical interventions that have been done under general anesthesia; they therefore have an increased probability to develop AKI.

N-acetylcysteine (NAC), a thiol compound with antioxidant and vasodilatory properties, reduces oxygen free radical production, decreases pump-related ischemia-reperfusion injury and the levels of pro-inflammatory cytokines. NAC has been reported to protect the kidney from injury induced by contrast media, ischemia, and toxins.

Present study aimed to explore the efficacy of NAC treatment to prevent deterioration in renal functioning in CKD patients undergoing major surgery under general anesthesia.

Study will include about 200 CKD (eGFR (estimated glomerular filtration rate) less than 40) patients that should undergo surgical interventions under general anesthesia and will divide to 3 groups as follows: group 1- about 40 patients which should undergo major vascular surgery; group 2 - about 60 patients that suppose to undergo major orthopedic surgery (revision of total hip, revision of knee); group 3 - about 100 patients undergoing major abdominal surgery. Patients from each group will randomly divide in two sub-groups (A and B). Subgroup A will receive NAC twice (14-16h and 2h) before surgery and 12h after surgery. Subgroup B will receive placebo (saline).

Markers for kidney function such as eGFR, creatinin, urea, electrolytes, cystatin C, NGAL (Neutrophil Gelatinase-Associated Lipocalin), urine albumin will measure before and after surgery in all patients. An additional blood samples for assessment of nitric oxide and cytokine levels will be taken from each patient before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from chronic kidney disease that should undergo surgical interventions under general anesthesia

Exclusion Criteria:

* pregnancy
* single kidney
* heart failure (NYHA class III-IV)
* hepatic failure
* mental diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2011-01; Primary Completion 2013-09 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
parameters of kidney function

CONTACTS AND LOCATIONS:
Overall Officials: Murat Bahar, MD, Study Chair — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel